CLINICAL TRIAL: NCT05298319
Title: The 90% Effective Flow of High Flow Nasal Oxygenation During Deeply Sedated Bronchoscopy
Brief Title: The 90% Effective Flow of High Flow Nasal Oxygenation (HFNO) During Sedated Bronchoscopy
Acronym: HFNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, attending, principle investigator, department of anesthesiology, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Zhejiang Cancer Hospital
Record Dates: First submitted 2022-02-28; First posted 2022-03-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia
Keywords: high flow nasal oxygenation; hypoxemia; bronchoscopy; effective flow
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): 10 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula
- Group 2 (Experimental): 20 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula
- Group 3 (Experimental): 30 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula
- Group 4 (Experimental): 40 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula
- Group 5 (Experimental): 50 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula
- Group 6 (Experimental): 60 L/min of oxygen flow
  Interventions: Device: high flow nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula — The patients were randomized into 6 groups, each group received different flow of oxygen, to observe the incidence of hypoxemia between different groups.

SUMMARY:
Patients undergoing sedated bronchoscopy were randomized into six groups (10 Liters/minute [L/min], 20 L/min, 30 L/min, 40 L/min, 50 L/min, 60 L/min). The primary outcome was the incidence of hypoxemia.

DETAILED DESCRIPTION:
It's a double-blind, randomized trial. The patients'demographic information, such as sex, weight, height, smoking status, present illness and history of past illness, were collected. After successful peripheral intravenous access, all patients, before sedation, received 20 min nebulization with lidocaine via a nebuliser facemask. The basic oxygen saturation, heart rate, and blood pressure of the patients were recorded by the investigators.Patients in the HFNO group received humidified oxygen at different rates via a high-flow nasal cannula (AIRVO2, New Zealand). After sedation with propofol and sufentanil, continuous electrocardiography and pulse oximetry were recorded, and the blood pressure of the patients was monitored throughout the procedure. . After bronchoscopy, patients were transferred to the post anesthesia care unit (PACU) if their vital signs were stable.

ELIGIBILITY:
Inclusion Criteria:

* (1) undergoing sedated bronchoscopy
* (2) 18 to 70 years of age;
* (3) American Society of Anaesthesiologists (ASA) class: I-III

Exclusion Criteria:

* (1) severe cardiac disease, including aortic stenosis, mitral stenosis, hemodynamic instability caused by severe arrhythmia, and acute myocardial infarction or cardiac surgery within the last 6 months;
* (2) severe hypoxemia (SpO2 < 90% without oxygen supply on admission), caused by interstitial lung disease, end-stage chronic obstructive pulmonary disease (COPD) or other diseases;
* (3) upper respiratory tract infection or lung infection;
* (4) refusal to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
the incidence of hypoxemia | during bronchoscopy
  hypoxemia was defined as SpO2 < 90%

SECONDARY OUTCOMES:
jaw thrust maneuver | during bronchoscopy
  percentage of jaw thrust maneuver
increase of flow rate | during bronchoscopy
  percentage of increase of flow rate
bag-mask ventilation | during bronchoscopy
  percentage of bag-mask ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang W, Yuan X, Shen Y, Wang J, Xie K, Chen X. Optimal flow of high-flow nasal cannula oxygenation to prevent desaturation during sedation for bronchoscopy: a randomized controlled study. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241246637. doi: 10.1177/17534666241246637. PMID 38659187